CLINICAL TRIAL: NCT04521231
Title: A Phase 1/2 Open-label Study to Investigate the Safety, Efficacy, and Pharmacokinetics of Administration of Subcutaneous Blinatumomab for the Treatment of Adults and Adolescents With Relapsed or Refractory B Cell Precursor Acute Lymphoblastic Leukemia (R/R B-ALL) and Minimal Residual Disease Positive (MRD+) B-ALL
Brief Title: A Study of Subcutaneous Blinatumomab Administration in Participants With R/R and MRD+ B-ALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20180257; 2023-506136-32 (EudraCT Number)
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: B Cell Precursor Acute Lymphoblastic Leukemia
Keywords: R/R B-ALL; MRD+ B-ALL; Relapsed; Refractory; Minimal Residual Disease; AMG 103; Blinatumomab; Acute lymphoblastic leukemia; Adolescent; Adult
MeSH Terms: conditions — Recurrence; Neoplasm, Residual; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation Phase: Blinatumomab Subcutaneous Formulation 1 (SC1) (Experimental): Cohorts of at least 3 adult participants with R/R B-ALL will be treated with escalating doses of blinatumomab to determine the maximum tolerated dose (MTD). The MTD will be defined as the dose for which the estimate of the toxicity rate from an isotonic regression (Yan et al, 2017) is closest to the target toxicity rate. Safety, pharmacokinetics (PK), pharmacodynamics (PD) and efficacy will be assessed.
  Interventions: Drug: Blinatumomab
- Dose Expansion Phase: Blinatumomab SC1 (Experimental): Up to 4 cohorts of adult participants with R/R B-ALL will be enrolled at different dose levels to support identification of the RP2D. Each cohort will aim to further assess safety, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy.
  Interventions: Drug: Blinatumomab
- Ph-IIC: Clinical PK Evaluation of SC Blinatumomab Formulations (Experimental): 1 cohort of adult participants will be enrolled into the Ph-IIC arm. The clinical PK evaluation cohort (Ph-IIC) will be conducted to compare the PK of SC1 and SC2 formulations at the preliminary RP2D determined from the dose expansion phase, in participants with R/R B-ALL.
  Interventions: Drug: Blinatumomab
- Ph-IIR: Efficacy of SC Blinatumomab in Participants with R/R B-ALL (Experimental): The efficacy of SC blinatumomab (in the SC2 formulation) will be evaluated in adults and adolescents with R/R B-ALL.
  Interventions: Drug: Blinatumomab
- Ph-IIM: Efficacy of SC Blinatumomab in Participants with MRD+ B-ALL (Experimental): The efficacy of SC blinatumomab (in the SC2 formulation) will be evaluated in adults and adolescents with MRD+ B-ALL.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab will be administered as a subcutaneous (SC) injection.
  Other Names: AMG 103

SUMMARY:
The Phase I part of the study aims to evaluate the safety, efficacy, and tolerability of subcutaneous (SC) blinatumomab for treatment of Relapsed or Refractory B cell Precursor Acute Lymphoblastic Leukemia (R/R B-ALL), to determine the maximum tolerated dose (MTD), and recommended phase 2 dose(s) (RP2D) of SC administered blinatumomab.

The Phase II part of the study will evaluate the safety, efficacy, and tolerability of SC blinatumomab for treatment of R/R B-ALL and Minimum Residual Disease Positive (MRD+) B-ALL in participants 12 years old and greater. It will also conduct a clinical pharmacokinetic (PK) evaluation of SC1 and SC2 blinatumomab formulations.

ELIGIBILITY:
Inclusion Criteria:

* Ph-IIC, Dose Escalation and Dose Expansion: Aged 18 years or older (or same or greater than legal age within the country if it is older than 18 years).
* Ph-IIRa and Ph-IIMa: Aged ≥ 17 years at time of informed consent.
* Ph-IIRb and Ph-IIMb: Age ≥ 12 years and < 17 years at time of informed consent.
* Ph-IIR, Ph-IIC, Dose escalation, Dose Expansion: Participants with R/R B-precursor ALL.
* Relapsed or Refractory B-precursor ALL at any time after first salvage therapy.
* Relapsed B-precursor ALL at any time after allogenic hematopoietic stem cell transplant (HSCT).
* Ph-IIR, Ph-IIC, Dose escalation, Dose expansion: Greater than or equal to 5% blasts in the Bone Marrow per local assessment.
* Ph-IIM: B-precursor ALL and bone marrow blasts (BMB) ≥ 0.01% and < 5% per local assessment.
* Ph-IIM: Availability of an appropriate archival BM specimen from initial or relapse diagnosis and the screening BM sample.
* Participants aged ≥ 18 years: Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2.
* Participants aged 16 to < 18 years old: Karnofsky Performance Score ≥ 50%.
* Participants aged < 16 years old: Lansky Performance Score ≥ 50%.
* Any Ph+ participant intolerant or refractory to prior tyrosine kinase inhibitors (TKIs) are eligible.
* Ph-IIM: BM function as follows:

  * Absolute Neutrophil Count (ANC) ≥ 500/μL
  * Platelet count ≥ 50 000/μL (transfusion permitted)
  * Hemoglobin level ≥ 9 g/dL (transfusion permitted)

The above is a summary, other inclusion criteria details may apply.

Exclusion Criteria:

* Active ALL in the central nervous system (CNS). Presence of greater than 5 white blood cells per cubic millimeter in cerebrospinal fluid (CSF) with lymphoblasts present and/or clinical signs of CNS leukemia. If CSF leukemia is present subjects will have to receive intrathecal therapy and have documented negative CSF prior to enrolling.
* History or presence of clinically relevant CNS pathology (excluding headache) such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis or severe (≥ grade 3) CNS events including immune effector cell-associated neurotoxicity syndrome (ICANS) from prior chimeric antigen receptor T-cell (CAR T) or other T cell engager therapies.
* Isolated Extramedullary (EM) Disease.
* For Ph-IIM only: Current EM disease or presence of circulating leukemia blasts.
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement.
* Active acute or chronic graft versus host disease requiring systemic treatment with immunosuppressive medication.
* Symptoms and/or signs that indicate an acute or uncontrolled chronic infection, any other disease or condition that could be exacerbated by the treatment or would complicate protocol compliance.
* Testicular leukemia.
* History of malignancy (with certain exceptions) other than ALL within 3 years prior to start of protocol-specified therapy.
* Allogeneic HSCT within 12 weeks before the start of protocol-specified therapy.
* Cancer chemotherapy within 2 weeks before the start of protocol-specified therapy (with certain exceptions).
* Immunotherapy within 4 weeks before start of protocol-specified therapy.
* Prior failed cluster of differentiation (CD19) directed therapy such as prior blinatumomab or CD19 CAR T cells will be allowed (with demonstrated continued CD19+ expression), if treatment ended more than 4 weeks prior to start of protocol therapy and no prior CNS complications.
* Currently receiving treatment in or less than 30 days or 5 half-lives since ending treatment on another investigational study(ies).
* Abnormal screening laboratory parameters.
* Female participant: Pregnant or breastfeeding or planning to become pregnant or donate eggs, or expected to breastfeed during treatment and for 96 hours after the last dose of investigational product (SC blinatumomab).

The above is a summary, other exclusion criteria details may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 281 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2027-11-24 (Estimated); Study Completion 2029-05-25 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Phase: Number of participants who experience dose limiting toxicities (DLTs) | Up to 29 days
Dose Escalation Phase: Number of participants who experience one or more treatment-emergent adverse events (TEAEs) | Up to approximately 28 weeks
Dose Escalation Phase: Number of participants who experience one or more serious TEAEs | Up to approximately 28 weeks
Dose Escalation Phase: Number of participants who experience one or more treatment-related TEAEs | Up to approximately 28 weeks
Dose Escalation Phase: Number of participants who experience one or more adverse events (AEs) of Interest (AEIs) | Up to approximately 28 weeks
Dose Expansion and Phase 2 Ph-IIR cohort: Number of participants who achieve complete remission (CR) / complete remission with partial hematological recovery (CRh) | Up to 10 weeks
Phase 2 Ph-IIC cohort: Maximum concentration (Cmax) of blinatumomab SC1 and SC2 | Up to approximately 4 weeks
Phase 2 Ph-IIC cohort: Average concentration (Cavg) of blinatumomab SC1 and SC2 | Up to approximately 4 weeks
Phase 2 Ph-IIC cohort: Time to reach maximum concentration (Tmax) of blinatumomab SC1 and SC2 | Up to approximately 4 weeks
Phase 2 Ph-IIC cohort: Area under the concentration-time curve (AUC) of blinatumomab SC1 and SC2 | Up to approximately 4 weeks
Phase 2 Ph-IIM cohort: Number of participants who achieve CR with MRD-negative response | Up to 10 weeks

SECONDARY OUTCOMES:
Dose Escalation and Dose Expansion Phase: Minimum concentration over the dosing interval (Cmin) of blinatumomab | Up to approximately 10 weeks
Dose Escalation and Dose Expansion Phase: Cmax of blinatumomab | Up to approximately 10 weeks
Dose Escalation and Dose Expansion Phase: Tmax of blinatumomab | Up to approximately 10 weeks
Dose Escalation and Dose Expansion Phase: AUC of blinatumomab | Up to approximately 10 weeks
Dose Escalation Phase and Phase 2 (Ph-IIC cohort): Number of participants who achieve CR/CRh | Up to 10 weeks
Dose Escalation Phase, Dose Expansion Phase and Phase 2 (Ph-IIR cohort, Ph-IIM cohort and Ph-IIC cohort): Number of participants with incidence of anti-blinatumomab antibody formation | Up to approximately 28 weeks
Dose Expansion Phase and Phase 2 (Ph-IIR cohort, Ph-IIM cohort and Ph-IIC cohort): Overall survival (OS) | Up to approximately 2 years
Dose Expansion Phase and Phase 2 (Ph-IIR cohort and Ph-IIC cohort): Duration of response | Up to approximately 2 years
Dose Expansion Phase and Phase 2 (Ph-IIR cohort, Ph-IIM cohort and Ph-IIC cohort): Relapse free survival | Up to approximately 2 years
Dose Expansion Phase and Phase 2 (Ph-IIR cohort, Ph-IIM cohort and Ph-IIC cohort): Number of participants who experience one or more TEAEs | Up to approximately 28 weeks
Dose Expansion Phase and Phase 2 (Ph-IIR cohort, Ph-IIM cohort and Ph-IIC cohort): Number of participants who experience one or more serious treatment-emergent adverse event | Up to approximately 2 years
Dose Expansion Phase and Phase 2 (Ph-IIR cohort, Ph-IIM cohort and Ph-IIC cohort): Number of participants who experience one or more treatment-related treatment-emergent adverse events | Up to approximately 28 weeks
Dose Expansion Phase and Phase 2 (Ph-IIR cohort, Ph-IIM cohort and Ph-IIC cohort): Number of participants who experience one or more AEIs | Up to approximately 28 weeks
Dose Expansion Phase and Phase 2 (Ph-IIR cohort, Ph-IIM cohort and Ph-IIC cohort): Summary scores of quality of life at each assessment as assessed by the EORTC QLQ-C30 for participants aged ≥ 17 years at the time of consent | Baseline (Day 1) up to approximately 28 weeks
  The EORTC QLQ-C30 is defined as the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire.
Dose Expansion Phase and Phase 2 (Ph-IIR cohort, Ph-IIM cohort and Ph-IIC cohort): Change from baseline of quality of life as assessed by the EORTC QLQ-C30 for participants aged ≥ 17 years at the time of consent | Baseline (Day 1) up to approximately 28 weeks
Phase 2 (Ph-IIR cohort and Ph-IIM cohort): Summary scores of quality of life at each assessment as assessed by PedsQL Generic Core Scale for participants aged 12 to < 17 years at time of consent | Baseline (Day 1) up to approximately 28 weeks
Phase 2 (Ph-IIR cohort and Ph-IIM cohort): Change from baseline of quality of life as assessed by PedsQL Generic Core Scale for participants aged 12 to < 17 years at time of consent | Baseline (Day 1) up to approximately 28 weeks
Phase 2 (Ph-IIR cohort): Number of participants who achieve CR | Up to 10 weeks
Phase 2 (Ph-IIR cohort): Number of participants who achieve CR, CRh, CRi (complete remission with incomplete hematological recovery) or blast free hypoplastic or aplastic bone marrow (BM) | Up to 10 weeks
Phase 2 (Ph-IIM cohort): Number of participants who achieve CR, CRh, CRi or blast free hypoplastic or aplastic BM with MRD-negative response | Up to 10 weeks
Phase 2 (Ph-IIR cohort and Ph-IIM cohort): Number of participants who achieve CR or CRh with MRD-negative response | Up to 10 weeks
Phase 2 (Ph-IIR cohort and Ph-IIM cohort): Duration of molecular response | Up to approximately 2 years
Phase 2 (Ph-IIR cohort and Ph-IIM cohort): Cmax of blinatumomab for participants participating in intense PK sampling assessment | Up to approximately 4 weeks
Phase 2 (Ph-IIR cohort and Ph-IIM cohort): Tmax of blinatumomab for participants participating in intense PK sampling assessment | Up to approximately 4 weeks
Phase 2 (Ph-IIR cohort and Ph-IIM cohort): AUC of blinatumomab for participants participating in intense PK sampling assessment | Up to approximately 4 weeks
Phase 2 (Ph-IIR cohort and Ph-IIM cohort): Blinatumomab serum concentrations for participants not participating in intense PK sampling assessment | Up to approximately 4 weeks
Phase 2 (Ph-IIR cohort and Ph-IIM cohort): Proportion of time on treatment with high side effect bother from baseline to end of treatment as measured by Functional Assessment of Chronic Illness Therapy (FACIT) GP5 item for participants aged ≥ 17 years | Baseline (Day 1) up to approximately 28 weeks
  This endpoint applies to participants aged ≥ 17 years at time of consent.
Phase 2 (Ph-IIR cohort and Ph-IIM cohort): Pain difference between pain score before and after injection as reported using the Numeric Rating Scale (NRS-11) for participants aged 12 to < 17 years at time of consent | Up to approximately 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (72):
- United States (9):
  - City of Hope National Medical Center, Duarte, California
  - University of Illinois Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - C.S. Mott Children's Hospital - University of Michigan, Ann Arbor, Michigan
  - New York University Grossman School of Medicine and New York University Langone Hospitals, New York, New York
  - Albert Einstein College of Medicine - Montefiore Medical Center, The Bronx, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - Sydney Childrens Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Queensland Childrens Hospital, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna, Austria
- Canada (4):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
- China (8):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Zhujiang Hospital of Southern Medical Unversity, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
- France (8):
  - Centre Hospitalier de Versailles - Hopital Andre Mignot, Le Chesnay
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Nice - Hopital de l Archet, Nice
  - Hopital Saint Louis, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Robert Debre, Paris
  - Hopital Lyon Sud, Pierre-Bénite
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
- Germany (8):
  - Universitaetsklinikum Augsburg, Augsburg
  - Charite - Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong
- Italy (7):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni xxiii, Bergamo
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant Orsola, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera di Rilievo Nazionale Santobono Pausilipon, Napoli
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
- Japan (5):
  - Akita University Hospital, Akita, Akita
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kanagawa Childrens Medical Center, Yokohami-shi, Kanagawa
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- South Korea (3):
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (8):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Complejo Asistencial Universitario de Salamanca Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Institut Catala d Oncologia Badalona Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Infantil Niño Jesus, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Turkey (Türkiye) (2):
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Izmir Ekonomi Universitesi Medical Point Hastanesi, Izmir

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Jabbour E, Zugmaier G, Agrawal V, Martinez-Sanchez P, Rifon Roca JJ, Cassaday RD, Boll B, Rijneveld A, Abdul-Hay M, Huguet F, Cluzeau T, Diaz MT, Vucinic V, Gonzalez-Campos J, Rambaldi A, Schwartz S, Berthon C, Hernandez-Rivas JM, Gordon PR, Bruggemann M, Hamidi A, Chen Y, Wong HL, Panwar B, Katlinskaya Y, Markovic A, Kantarjian H. Single agent subcutaneous blinatumomab for advanced acute lymphoblastic leukemia. Am J Hematol. 2024 Apr;99(4):586-595. doi: 10.1002/ajh.27227. Epub 2024 Feb 5. PMID 38317420
- [Derived] Jabbour E, Lussana F, Martinez-Sanchez P, Torrent A, Rifon JJ, Agrawal V, Tormo M, Cassaday RD, Cluzeau T, Huguet F, Papayannidis C, Hernandez-Rivas JM, Rijneveld A, Fleming S, Vucinic V, Boll B, Ikezoe T, Abdul-Hay M, Savoie ML, Schuh AC, Berthon C, Schwartz S, Chiaretti S, Yuda J, Miyazaki T, Gonzalez-Campos J, Chen Y, Wong H, Choudhry J, Zugmaier G, Guest E, Gordon P, Kantarjian H. Subcutaneous blinatumomab in adults with relapsed or refractory B-cell acute lymphoblastic leukaemia: post-hoc safety and activity analysis from a multicentre, single-arm, phase 1/2 trial. Lancet Haematol. 2025 Jul;12(7):e529-e541. doi: 10.1016/S2352-3026(25)00144-9. Epub 2025 Jun 15. PMID 40532723
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com